CLINICAL TRIAL: NCT06717646
Title: Laser Spatiotemporal Photoplethysmogram and Computational Method for Extended Chronic Cardiometabolic Therapeutic Care
Brief Title: Using Laser Spatiotemporal Photoplethysmogram and Computational Method for Management of Chronic Disorders.
Acronym: LSPPG
Status: Recruiting | Type: Observational
Sponsor: National Heart Centre Singapore (Other)
Collaborators: National Medical Research Council (NMRC), Singapore (Other Government)
Responsible Party: Sponsor
Other Study IDs: 2021/2724
Record Dates: First submitted 2024-11-18; First posted 2024-12-05 (Actual); Last update posted 2024-12-05 (Actual); Status verified 2024-03

CONDITIONS: Blood Glucose Monitoring; Blood Pressure Measurement

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Inpatient: Patients warded under National Heart Centre Singapore
- Outpatients: Patients scheduled for 24-hour Ambulatory Blood Pressure Monitoring at National Heart Centre Singapore

SUMMARY:
This investigational study is carried out to find out if a smartwatch monitor worn on the wrist that acts like a blood pressure monitor, will be able to replace the traditional blood pressure measurements using the traditional cuff that is wrapped around your arm.

DETAILED DESCRIPTION:
NHC inpatients (Group A) Patients will be required to put on the LSPPG wearable sensor to take measurement once a day, starting from the day of recruitment till day of discharge. 3 ECG electrodes with cable linking to the LSPPG sensor wearable will also be attached on the chest. This helps to capture ECG rhythm at the same time. Study team member will assist the patient to take daily measurement.

NHC Outpatients scheduled for 24-Hour ABP monitoring (Group B) Patients will wear the LSPPG wearable sensor whilst wearing the 24-hour ambulatory blood pressure monitor. 3 ECG electrodes with cable linking to the LSPPG sensor wearable will also be attached on the chest. This helps to capture ECG rhythm at the same time. Readings will be obtained on an hourly basis during the duration of wearing the ambulatory blood pressure machine (clinical grade device).

ELIGIBILITY:
Inclusion Criteria:

* Above 21 years of age
* Sufficient language skills in English, Chinese, Malay or Tamil
* Provided informed consent

Exclusion Criteria:

* Skin sensitivity to adhesives

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients from National Heart Centre Singapore
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2024-04-11 (Actual); Primary Completion 2025-06 (Estimated); Study Completion 2025-06 (Estimated)

PRIMARY OUTCOMES:
Comparable results to traditional methods | 24 Hours
  Perform comparably to the 24-hour ambulatory blood pressure meters and continuous glucose monitors (CGM) to establish hypertension and blood glucose changes
Improve efficiency | 24 Hours
  Provide real time feedback to patients and healthcare providers to individualize hypertension / hyperglycemic treatment
Lifestyle Improvement | 24 Hours
  Consider patient lifestyle changes and reduce medication burden, especially in the elderly when blood pressure control is optimal.

CONTACTS AND LOCATIONS:
Locations (1):
- National Heart Centre Singapore, Singapore, Singapore

IPD SHARING:
Plan to Share IPD: Yes